CLINICAL TRIAL: NCT07148609
Title: Video Game-facilitated Group Activity for Quality of Life and Social Function in Chronic Schizophrenia Inpatients: A Randomized Controlled Parallel-group Pilot Trial.
Brief Title: Video Game-facilitated Group Activity for Quality of Life and Social Function in Chronic Schizophrenia Inpatients.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Principal Investigator, Wei-Yu Chiang, Resident psychiatrist, TsaoTun Psychiatric Center, Department of Health, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TTPC-114015
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Patients
Keywords: Video game; Schizophrenia; Social function; Quality of life
MeSH Terms: conditions — Schizophrenia; Social Adjustment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Active Comparator)
  Interventions: Behavioral: Video game-facilitated group activity
- Controlled arm (No Intervention)

INTERVENTIONS:
Behavioral: Video game-facilitated group activity — The intervention is a 12-week group activity program for each participant in the intervention group, and the program consists of three 50-minute video game facilitated group activity sessions per week. Participants in the intervention group will engage in those group activity session which will be mediated by the game of Super Mario Party on Nintendo Switch.
  Arms: Interventional arm

SUMMARY:
The goal of this clinical trial is to learn if video game-facilitated group activity helps to improve the quality of life and social function in inpatients with chronic schizophrenia.

The main questions it aims to answer are:

* Does video game-facilitated group activity enhance the quality of life as measured by a standardized scale (WHOQOL) in patients with schizophrenia hospitalized in a psychiatric hospital?
* Can video game-facilitated group activity promote social function as measured by a specific scale (PSP) in patients with schizophrenia hospitalized in a psychiatric hospital?

Researchers will compare video game-facilitated group activity to regular occupational therapy to see if the intervention is beneficial to patients with chronic schizophrenia.

Participants will:

* Attend to video game-facilitated group activity or regular occupational therapy three times a week for 12 weeks.
* Receive assessments upon and after the 12-week intervention, and another 12 weeks after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between >18 and <65 years with a principal diagnosis of schizophrenia, as defined by the International Classification of Diseases (ICD-10) codes F20.0-F20.9 which was diagnosed according to DSM-5-TR criteria.
* Possessing a valid Catastrophic Illness Certificate for schizophrenia and being continuously hospitalized for more than six months.
* Being able to read Chinese and communicate effectively in either Mandarin or Taiwanese.
* Being able to comprehend the purpose of the study and to provide written informed consent after the study has been explained by the researchers.

Exclusion Criteria:

* Individuals exhibiting unstable psychiatric or consciousness conditions, or those unable to comply with video game-based instruction and operation.
* Individuals with a history of ocular diseases, severe cardiovascular disorders, epilepsy, or brain injuries; or those who have experienced acute cardiovascular or cerebrovascular events, bone fractures, undergone hip or knee joint replacement, or present with lower limb balance impairments or structural injuries-such as amputations, post-lumbar surgery status, or acute ankle sprains-rendering participation unsuitable within the past six months.
* Concurrent participation in other research studies during the study period, where the intervention may potentially influence the primary or secondary outcomes of this study.
* Individuals who are legally declared under guardianship.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The changes of quality of life | The outcome will be assessed at baseline, week 12, and week 24.
  The changes of quality of life will be assessed by the World Health Organization Quality of Life-BREF (WHOQOL-BREF).
The changes of social function. | The outcome will be assessed at baseline, week 12, and week 24
  The changes of social function will be evaluated by the Personal and Social Performance Scale (PSP).

SECONDARY OUTCOMES:
The changes of cerebral blood flow. | The outcome will be assessed at baseline and week 12.
  The changes in cerebral blood be measured by Near-Infrared Spectroscopy (NIRS).
The change of cognitive function. | The outcome will be assessed at baseline and week 12.
  The Montreal Cognitive Assessment (MoCA) will be used to evaluate changes in cognitive function.
The change of psychiatric symptoms. | The outcome will be assessed at baseline and week 12.
  The Brief Psychiatric Rating Scale (BPRS) will be used to assess changes in positive and negative psychiatric symptoms.
The change of physical fitness | The outcome will be assessed at baseline and week 12.
  Physical fitness assessments will be conducted to measure changes in participants' physical fitness levels, including cardiopulmonary endurance, the strength and flexibility of upper and lower limbs, as well as dynamic and static balance.
  * The cardiopulmonary endurance would be measured by 6-minute walk test and march-in-place test.
  * The upper limbs strength will be measured by arm curl test and hand grip strength test.
  * The lower limbs strength will be measured by 30-second chair stand test.
  * The upper limbs flexibility will be measured by back scratch test.
  * The lower limbs flexibility will be measured by chair sit-and-reach test.
  * The dynamic balance test will be measured by chair stand and obstacle walk test.
  * The static balance test will be measured by one-leg stand test with eyes open.

OTHER OUTCOMES:
Demographic data | Demographic data will be assessed at baseline.
  Demographic data including age, sex, marital status, educational year, body mass index, past medical and allergic history, and other information related with this study will be assessed by research assistants.
The change of daily antipsychotic dose equivalences. | This outcome will be assessed at the baseline, Week 12, and Week 24.
  The dosage of antipsychotic medications of the participants will be calculated according to their usage of antipsychotic medications that are equivalent to 100 mg/day of chlorpromazine. The daily antipsychotic dose equivalences will be calculated by the average of the daily dose equivalences in the weeks that are scheduled to be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jen Yang, Study Chair — Tsao-Tun Psychiatric Center
Locations (1):
- Tsao-Tun Psychiatric Center, Ministry of Health and Welfare, Nantou City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No